CLINICAL TRIAL: NCT01577485
Title: LGG/BB12-pastille Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of Michigan (Other); The Forsyth Institute (Other)
Responsible Party: Principal Investigator, Eva Soderling, Associate Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: ETMK:22/180/2012
Record Dates: First submitted 2012-04-12; First posted 2012-04-13 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Probiotics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic pastille (Experimental): Test group
  Interventions: Dietary Supplement: Probiotics in an pastille
- Control pastille (Active Comparator): Control group
  Interventions: Dietary Supplement: Control pastille

INTERVENTIONS:
Dietary Supplement: Probiotics in an pastille — Test group
  Arms: Probiotic pastille
Dietary Supplement: Control pastille — Control group
  Arms: Control pastille

SUMMARY:
We want to study the effect of short-term consumption of probiotics (a mixture of L. rhamnosus GG and B. lactis BB-12)on the composition of the oral flora.

ELIGIBILITY:
Inclusion Criteria:

* Subjects healthy, 20-30 yrs of age

Exclusion Criteria:

* Subjects not healthy, too old/young

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Counts of mutans streptococci | 4 weeks

SECONDARY OUTCOMES:
Amount of plaque | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Söderling, Principal Investigator — Associate Professor
Locations (1):
- Institute of Dentistry, Turku, Finland